CLINICAL TRIAL: NCT01562301
Title: A Phase I Study of the Combination of Carboplatin, Docetaxel, and Increasing Doses of Sublingual Anvirzel (Nerium Oleander) in Advance Non-Small Cell Lung Cancer
Brief Title: Sublingual Anvirzel in Advance Non-Small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Nerium Biotechnology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0147; MDA-2011-0147; CDR0000728644 (Other: NCI Clinical Trials); NCI-2012-00709 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Chemotherapeutic Agent Toxicity; Lung Cancer
Keywords: chemotherapeutic agent toxicity; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; carboplatin; Paraplatin; docetaxel; Taxotere; Anvirzel; nerium oleander; Advanced Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Docetaxel; Anvirzel; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anvirzel + Carboplatin + Docetaxel (Experimental): Anvirzel administered sublingually. A total of five dose cohorts evaluated (6, 12, 24, 36, 48 mg/m2/day; SL divided into 3 doses given every 8 hrs) with 3 patients per cohort. Patients receive the assigned dose (2, 4, 8, 12, or 16 mg/m2) of Anvirzel three times a day throughout each cycle for a total of 4 cycles of chemotherapy. Cycles occur every 21 days. Patients start with an AUC of 6 for Carboplatin and 75mg/m2 for docetaxel, and on subsequent cycles, modifications at the discretion of the treating team. Questionnaire completion regarding physical and mental at baseline, 7 days before chemotherapy, day 1 of chemotherapy, day 1 of cycles 2, 3, and 4, and at end of dosing visit.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Drug: Anvirzel; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Carboplatin — AUC 6 by vein 7 days after Anvirzel administration in a 21 dayc cycle.
  Other Names: Paraplatin
Drug: Docetaxel — 75 mg/m2 by vein 7 days after Anvirzel administration in a 21 day cycle.
  Other Names: Taxotere
Drug: Anvirzel — Starting Cohort Dose: 6 mg/m2 given 3 times a day administered sublingually for a 21 day cycle.
  Expansion Cohort Starting Dose: Maximum tolerated dose from
  Other Names: Nerium oleander
Behavioral: Questionnaires — Questionnaire completion regarding physical and mental at baseline, 7 days before chemotherapy, day 1 of chemotherapy, day 1 of cycles 2, 3, and 4, and at end of dosing visit.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Anvirzel (Nerium Oleander) that can be given to lung cancer patients receiving standard therapy with carboplatin and docetaxel. Researchers also want to learn what effect Nerium Oleander may have in combination with carboplatin and docetaxel.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are eligible and agree to take part in the study, you will be assigned to a dose level of nerium oleander based on when you join this study. Up to 5 dose levels of nerium oleander will be tested. At least 3 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of nerium oleander is found.

You will take nerium oleander by mouth by placing it under your tongue. You should hold the nerium oleander under your tongue for 3 minutes before swallowing. It is very important for you to hold the nerium oleander under your tongue for 3 full minutes. Holding it under your tongue for 3 minutes before swallowing helps your body to take in the highest amount of the drug that you can receive. If you hold the nerium oleander under your tongue for less than 3 minutes, your body will not receive as much of the study drug and may not possibly benefit as much. You will take nerium oleander 3 times a day while participating in this study. Nerium oleander should be taken on an empty stomach or at least 15 minutes before any large meal, to help your body take in as much of the drug as possible.

Study Visits:

Each of your chemotherapy cycles are 21 days.

Each week while on study, you will complete the questionnaire about any symptoms you may be having. It should take about 5 minutes to complete it each time.

Cycle 1:

On Day -7 (7 days before you start chemotherapy):

* You will complete the questionnaire about your physical and mental health. It should take about 5 minutes to complete it.
* Blood (about 2 teaspoons each time) will be drawn 6 times over 8 hours for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.
* Blood (about 6 teaspoons) will be drawn to learn if the study drug is reducing inflammation.
* Blood (about 2 teaspoons) will be drawn to test the effect of the study drug on your immune system.

On Day -6, blood (about 2 teaspoons each time) will be drawn 1 time for PK testing.

On Day 1 (the day you start chemotherapy):

* You will be asked about any symptoms you may be having or drugs you may be taking.
* You will have a physical exam, including measurement of weight and vital signs.
* Your performance status will be recorded.
* You will complete the questionnaire about your physical and mental health.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Blood (about 2 teaspoons each time) will be drawn 6 times over 8 hours for PK testing.
* Blood (about 6 teaspoons) will be drawn to learn if the study drug is reducing inflammation.
* Blood (about 2 teaspoons) will be drawn to test the effect of the study drug on your immune system.
* You will have an EKG.

On Day 2:

* Blood (about 2 teaspoons) will be drawn for PK testing.
* Blood (about 6 teaspoons) will be drawn to learn if the study drug is reducing inflammation.
* Blood (about 2 teaspoons) will be drawn to test the effect of the study drug on your immune system.

On Day 8 (+/- 2 days):

* Blood (about 6 teaspoons) will be drawn to learn if the study drug is reducing inflammation.
* Blood (about 2 teaspoons) will be drawn to test the effect of the study drug on your immune system.

On Day 1 of Cycles 2-3:

* You will be asked about any symptoms you may be having or drugs you may be taking.
* You will have a physical exam, including measurement of weight and vital signs.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Your performance status will be recorded.
* You will have an EKG.
* You will complete the questionnaire about your physical and mental health.
* On Day 1 of Cycle 3 only, you will have a CT scan to check the status of the disease.

On Day 1 of Cycle 4:

* You will be asked about any symptoms you may be having or drugs you may be taking.
* You will have a physical exam, including measurement of weight and vital signs.
* You will complete the questionnaire about your physical and mental health.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* Your performance status will be recorded.
* You will have an EKG.
* Blood (about 2 teaspoons each time) will be drawn 6 times over 8 hours for PK testing.
* Blood (about 6 teaspoons) will be drawn to learn if the study drug is reducing inflammation.
* Blood (about 2 teaspoons) will be drawn to test the effect of the study drug on your immune system.

On Day 2 of Cycle 4:

* Blood (about 2 teaspoons) will be drawn for PK testing.

On Day 8 and Day 21 of Cycle 4 (+/- 2 days):

* Blood (about 6 teaspoons) will be drawn to learn if the study drug is reducing inflammation.
* Blood (about 2 teaspoons) will be drawn to test the effect of the study drug on your immune system.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest or up to 4 cycles. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visit.

End-of-Dosing Visit:

After your last dose of study drug, you will return to the clinic. The following tests and procedures will be performed:

* You will be asked about any symptoms you may be having or drugs you may be taking.
* You will have a physical exam, including measurement of weight and vital signs.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will have an EKG.
* You will have a CT scan to check the status of the disease.
* You will complete both questionnaires.

Follow-Up Visit:

About 30 days after your last dose of study drug, the following tests and procedures will be performed:

* You will be asked about any symptoms you may be having or drugs you may be taking.
* You will have a physical exam, including measurement of weight and vital signs.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will have an EKG.
* You will complete both questionnaires.

This is an investigational study. Nerium oleander is not FDA approved or commercially available. Its use in this study is considered investigational.

Up to 36 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed diagnosed advanced non-small cell lung cancer (Stage IIIB and IV) and be scheduled to receive four cycles of carboplatin and docetaxel chemotherapy.
2. Newly diagnosed or previously treated patient with NSCLC. Previously treated patients are allowed to have any previous chemotherapy for the treatment of NSCLC.
3. Age >18 years
4. ECOG performance status < or =2 (Karnofsky > or = 60%)
5. Life expectancy of greater than 6 months
6. Patients must have normal organ and marrow function as defined below: - leukocytes > or = 3,000/mcL - absolute neutrophil count > or = 1,500/mcL - platelets > or = 100,000/mcL - total bilirubin within normal institutional limits - AST(SGOT)/ALT(SGPT) < or = 2.5 X institutional upper limit of normal - creatinine within normal institutional limits OR - creatinine clearance > or = 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
7. Negative serum or urine pregnancy test in women of child-bearing potential
8. Scheduled to begin carboplatin and docetaxel chemotherapy in the next 30 days
9. The effects of Anvirzel on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients receiving any other investigational agents
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cardiac glycosides
3. Patients receiving any medications or substances that are inhibitors or inducers of CYP 3A4 are ineligible
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant or breastfeeding women
6. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Anvirzel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
7. Uncontrolled or significant cardiovascular disease, including: • Myocardial infarction within 6 months • Uncontrolled angina within 6 months • Newly diagnosed congestive heart failure within 6 months, defined as NYHC-II or currently uncontrolled congestive heart failure • Diagnosed or suspected congenital long QT syndrome • Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, Wolff-Parkinson-White (WPW) syndrome, or torsade de pointes). Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec). If the automated reading is prolonged (i.e., > 450 msec), the EKG should be manually over-read • Any history of second or third degree heart block • Heart rate < 50 beats/minute or sustained heart rate > 110 on pre-entry electrocardiogram • Newly diagnosed atrial fibrillation within 6 months or currently uncontrolled atrial fibrillation • Uncontrolled hypertension defined as sustained blood pressure of >/= 140/90mm Hg
8. Current use of a pacemaker
9. Patients using or scheduled to use bevacizumab during study period
10. Current use of cardiac glycoside

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of sublingual (SL) dosing of Anvirzel in combination with chemotherapy | 21 Day Cycle
Pharmacokinetics of carboplatin and docetaxel when administered concurrently with SL Anvirzel | 24 hours
  Pharmacokinetic studies evaluate plasma concentrations over a 24 hour period prior to administration of chemotherapy, using high performance liquid chromatographic and electron ion-spray mass spectrometry

SECONDARY OUTCOMES:
Anti-inflammatory effects of SL Anvirzel during carboplatin and docetaxel chemotherapy | Up to four 21 day cycles (84 days)
Immunomodulatory effects of SL Anvirzel during carboplatin and docetaxel chemotherapy | Up to four 21 day cycles (84 days)
Symptoms and quality-of-life outcomes based on MDASI-LC and SF-12 scores | Up to four 21 day cycles (84 days)
Grade 3-4 toxicities at each course according to NCI Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0 | Up to four 21 day cycles (84 days)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Lee, MD, FACP, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org